CLINICAL TRIAL: NCT00486798
Title: FAST-A Study to Evaluate the Efficacy and Safety of Quetiapin IR in Patients With Acute Psychosis
Acronym: FAST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: study was not ethically acceptable to continue and therefore it was finally stopped
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00009; EUDRAC No. 2006-006426-26
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2009-04

CONDITIONS: Psychotic Disorders; Schizophrenia; Bipolar Disorder
Keywords: acute schizophrenia; schizoaffective disorder; psychosis Not Otherwise Specified (NOS); bipolar mania with psychotic symptoms
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder | interventions — Quetiapine Fumarate; Blood Specimen Collection

INTERVENTIONS:
Drug: Quetiapine
Procedure: Rating Scales
Procedure: Self Assessment Form
Procedure: Blood and urine samples
Procedure: Sleeping pattern

SUMMARY:
The purpose of this study is to compare the efficacy of quetiapine IR, following rapid titration versus conventional titration in patients with acute psychosis

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent
* male or female, aged 18-65 years
* requirement of hospitalization and in need for antipsychotic treatment for an acute psychotic episode
* able to swallow tablets from Day 1

Exclusion Criteria:

* In-patients who are anticipated to be discharged before evaluation of the primary outcome variable at Day 5
* patients with known relevant clinical disease
* history of syncope, or orthostatic hypotension
* patients with known neutropenia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Positive and Negative Syndrome Scale-Excitatory Subscale (PANSS-EC) at day 5 compared with baseline at day 1

SECONDARY OUTCOMES:
Assessment of PANSS-EC at Day 3 and 8. Clinical Global Impression (CGI) at baseline and at Day 5 and 8. FAST (For Acute Seroquel Therapy) rating scale at baseline and at Day 5 and 8. The sleeping pattern (8days). Withdrawals/treatment failures. AE

CONTACTS AND LOCATIONS:
Overall Officials: Jaan Ruusa, MD,PhD, Principal Investigator — Huddinge Hospital Stockholm Sweden; Birgit Ekholm, MD, Study Director — AstraZeneca Sweden AB
Locations (13):
- Sweden (13):
  - Research Site, Borås
  - Research Site, Danderyd
  - Research Site, Falköping
  - Research Site, Gothenburg
  - Research Site, Karlskrona
  - Research Site, Malmo
  - Research Site, Öjebyn
  - Research Site, Piteå
  - Research Site, Simrishamn
  - Research Site, Stockholm
  - Research Site, Trollhättan
  - Research Site, Vaxjo
  - Research Site, Västerås